CLINICAL TRIAL: NCT00316550
Title: A Randomized, Double-Blind, Placebo-Controlled, Cross-Over Pilot Study to Assess the Effects of AV608 on Central Processing of Visceral Stimuli in Subjects With Irritable Bowel Syndrome
Brief Title: Pilot Study to Assess the Effects of AV608 on Irritable Bowel Syndrome
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Animal Safety Data
Sponsor: Avera Pharmaceuticals (Industry)
Collaborators: University of California, Los Angeles (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AV608-107
Record Dates: First submitted 2006-04-19; First posted 2006-04-21 (Estimated); Last update posted 2008-02-25 (Estimated); Status verified 2008-02

CONDITIONS: Irritable Bowel Syndrome (IBS)
Keywords: Irritable Bowel Syndrome (IBS)
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: AV608

SUMMARY:
The purpose of this study is to assess the effects of AV608, a neurokinin 1 (NK-1) antagonist, in subjects with Irritable Bowel Syndrome.

DETAILED DESCRIPTION:
This is a single-center, randomized, double-blind, placebo-controlled, cross-over study to assess the effects of AV608 on brain processing of visceral stimuli and emotional visual cues in subjects with IBS. Female subjects between 18 and 65 years of age who meet diagnostic criteria for Irritable Bowel Syndrome will be eligible for the study.

Eligible subjects will complete a baseline fMRI imaging procedure that includes both emotional visual cues and visceral stimulation. All subjects who participate in the study will receive 3 weeks of treatment with AV608 and 3 weeks of treatment with placebo during the course of the study; the order of the two treatments for each subject will be randomly determined.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18 to 65 years of age, inclusive
* Current diagnosis of Irritable Bowel Syndrome (IBS)
* Subjects 50 years of age or older must have had a barium enema and flexible sigmoidoscopy or a colonoscopy and provide a record of this test
* Willing to participate in this study as evidenced by a signed, written informed consent form (ICF)
* If female and of child-bearing potential, willing to avoid pregnancy and practice adequate birth control from the time of study enrollment through at least 30 days after the final dose of study medication
* If female, negative pregnancy test results
* Right handed
* Ambulatory outpatient
* Agrees to refrain from blood donation during the course of the study
* Written and oral fluency in the English language

Exclusion Criteria:

* Evidence of structural abnormality of the gastrointestinal tract or GI diseases/conditions
* Current evidence or diagnosis of peptic ulcer
* Endoscopic bowel evaluation with evidence of cancer, inflammatory bowel disease, or other structural disease
* History of abdominal surgery such as adhesion lysis or any gastrointestinal surgery
* History of gastroesophageal reflux disease not controlled by a stable dose of medication
* Any evidence of or treatment of malignancy within the previous 5 years
* Clinical evidence of any disease that may interfere with participation in the study
* Existence of surgical or medical conditions which interfere with the absorption, distribution, metabolism and excretion of the study drug
* Symptoms of a significant clinical illness within the 2 weeks prior to Screening
* Type 1 diabetes mellitus, insulin-dependent Type 2 diabetes mellitus, and thyroid disorders or other endocrine disorders that are not well controlled by appropriate therapy
* A QTc interval of greater than or equal to 450 msec at Screening
* Presence of a psychotic disorder, bipolar disorder, alcohol or substance dependence (other than nicotine dependence) or eating disorder within the previous year according to DSM-IV-TR criteria
* Seizure disorder
* Subjects who have previously participated in a clinical trial for AV608 (previously known as NKP608 and CGP608)
* Positive drug test result at Screening
* Use of investigational drugs, products or devices within 30 days prior to Screening
* Planned use of certain drugs during the study that affect the central nervous system, gastrointestinal motility, autonomic activity or pain sensation
* Use of pimozide, terfenadine, astemizole, or cisapride during the study
* Presence of moderate or severe allergy
* Regular intake of more than 2 units of alcohol per day
* Pregnant or breast feeding
* Subjects with morbid obesity
* Subjects with metal implants or large tattoo
* Any clinically significant abnormalities on the Screening physical examination, ECG or laboratory tests
* Members of the investigative staff or their immediate family members
* Any other condition that the investigator believes would jeopardize the safety or rights of the subject or would render the subject unable to comply with the study protocol
* Regular use of more than 10 cigarettes per day

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2006-04; Primary Completion 2007-06 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the effect of AV608 on regional brain responses as measured by fMRI during conditioned and unconditioned visceral pain due to rectal distension.

SECONDARY OUTCOMES:
The effect of AV608 on regional brain responses to emotional visceral cues as measured by fMRI and the visceral pain threshold during rectal distension will be evaluated as secondary efficacy endpoints.

CONTACTS AND LOCATIONS:
Overall Officials: Joao Siffert, MD, Study Director — Avera Pharmaceuticals, Inc.; Kirsten Tillisch, MD, Principal Investigator — UCLA Center for Neurovisceral Sciences and Women's Health
Locations (1):
- UCLA Center for Neurovisceral Sciences and Women's Health, Los Angeles, California, United States